CLINICAL TRIAL: NCT04034745
Title: IIT2018-26 -Hendifar-NETCx: A Descriptive, Multicenter, Single-arm, Open Label Study to Analyze the Effect of Telotristat Ethyl on Weight Regulation/Gain
Brief Title: Open Label Study to Analyze the Effect of Telotristat Ethyl on Weight Regulation/Gain
Status: Withdrawn | Type: Observational
Why Stopped: lack of funding
Sponsor: Andrew Hendifar, MD (Other)
Collaborators: Lexicon Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Andrew Hendifar, MD, Assistant Professor of Medicine, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Other Study IDs: IIT2018-26 -Hendifar-NETCx
Record Dates: First submitted 2019-06-29; First posted 2019-07-26 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Pancreatic Cancer; Neuroendocrine Tumors; Cachexia; Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Neuroendocrine Tumors; Cachexia; Neoplasms | interventions — telotristat ethyl

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Standard of Care telotristat ethyl (Xermelo) Treatment: Treatment of telotristat ethyl (Xermelo) with DXA scans and bionutritional assessments (24-hour food recall and taste/smell alteration) conducted 3x during telotristat ethyl treatment.
  Interventions: Drug: telotristat ethyl

INTERVENTIONS:
Drug: telotristat ethyl — 250 mg tablets of Xermelo (telotristat ethyl) is administered orally 3x daily in combination with somatostatin analogs (SSAs) for approximately 84 days as per standard of care
  Other Names: Xermelo

SUMMARY:
This single arm study will evaluate whether Xermelo (telotristat ethyl) associated weight gain is affects lean body mass, dietary intake, and physical and cognitive functioning among neuroendocrine tumor (NET) patients with a history of carcinoid syndrome.

DETAILED DESCRIPTION:
The purpose of this study is to examine the mechanisms of weight gain associated with the drug telotristat ethyl (Xermelo) among patients with a neuroendocrine tumor (NET) with history of carcinoid syndrome. We want to know if taking Xermelo affects patients' lean body mass, quality of life, dietary intake, and physical and cognitive functioning during treatment. A better understanding of the mechanisms of weight gain from Xermelo may allow us to determine whether this drug may be beneficial for treating carcinoid syndrome, cachexia, or weight loss seen in other diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histopathologically confirmed diagnosis of a metastatic NET.
* Documented history of carcinoid syndrome.
* Currently receiving treatment with long-acting SSAs with a plan to initiate therapy with telotristat-ethyl as per standard of care.
* ECOG performance status 0-1 and/or Karnofsky >60%.
* Greater than or equal to 3 month life expectancy.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients experiencing more than 12 watery BMs per day associated with volume contraction, dehydration, or hypotension, or showing evidence of enteric infection.
* History of short bowel syndrome.
* Clinically important baseline elevation in liver function tests.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Malignant ascites requiring paracenteses.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Bowel obstruction, partial, or total.
* Pregnancy
* Patients with unresolved grade 3/4 adverse effects of prior therapy at time of enrollment, other than diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from Cedars-Sinai Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Mean change in lean body mass (measured using DXA Scan) from baseline and after 13 weeks of treatment. | From baseline to 13 weeks after treatment

SECONDARY OUTCOMES:
Mean change in patient reported outcomes using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) from baseline up to 3 years post treatment. | From baseline to 3 years post treatment
  The summary score (SS) is a mean of 13 QLQ-C30 subscale scores, ranging from 0 to 100, with a higher SS rating reflecting a better health status.
Mean change in patient reported outcomes using the Montreal Cognitive Assessment (MOCA) test from baseline up to 3 years post treatment. | From baseline to 3 years post treatment
  MOCA scores range between 0 and 30, with higher scores indicating higher cognitive function.
Mean change in patient reported outcomes using a stool survey measured from baseline and after 13 weeks of treatment. | From baseline to 13 weeks post-treatment.
  The stool survey is a non-validated descriptive measure of gastrointestinal symptoms by taking the mean score on a scale of 0 - 10, where 0 indicates no symptoms and higher scores denote a worsening of symptoms.
Mean change in calories consumed using a 24-hour food diary from baseline and after 13 weeks of treatment. | From baseline to 13 weeks post-treatment
Mean change in daily activity levels (steps) as measured using a wrist-worn fitness tracker (e.g., Fitbit) from baseline and for the duration of the 13 weeks of treatment. | From baseline to 13 weeks post-treatment
Mean change in daily activity levels [stairs (floors) climbed] as measured using a wrist-worn fitness tracker (e.g., Fitbit) from baseline and for the duration of the 13 weeks of treatment. | From baseline to 13 weeks post-treatment
Mean change in daily activity levels (sleep duration) as measured using a wrist-worn fitness tracker (e.g., Fitbit) from baseline and for the duration of the 13 weeks of treatment. | From baseline to 13 weeks post-treatment
Mean change in daily activity levels (heart rate) as measured using a wrist-worn fitness tracker (e.g., Fitbit) from baseline and for the duration of the 13 weeks of treatment. | From baseline to 13 weeks post-treatment
Mean change in daily activity levels (active minutes) as measured using a wrist-worn fitness tracker (e.g., Fitbit) from baseline and for the duration of the 13 weeks of treatment. | From baseline to 13 weeks post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Hendifar, MD, MPH, Principal Investigator — Cedars-Sinai Medical Center